CLINICAL TRIAL: NCT00084019
Title: A Prospective, Open-Label, Pilot Trial of Regimen Simplification to Atazanavir/Ritonavir Alone as Maintenance Antiretroviral Therapy After Sustained Virologic Suppression
Brief Title: Atazanavir/Ritonavir Maintenance Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A5201; 10096 (Registry Identifier: DAIDS ES); ACTG A5201
Record Dates: First submitted 2004-06-04; First posted 2004-06-07 (Estimated); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Treatment Experienced
MeSH Terms: conditions — HIV Infections | interventions — Atazanavir Sulfate; Ritonavir

INTERVENTIONS:
Drug: Atazanavir
Drug: Ritonavir

SUMMARY:
Long-term side effects, the expense of medications, and the difficulty of taking medications continuously for long periods of time are all problems with complicated anti-HIV drug regimens. The purpose of this study is to determine whether two drugs, atazanavir (ATV) and ritonavir (RTV), will control HIV infection when taken together without any other anti-HIV drugs after 48 weeks of viral suppression.

Hypothesis: Simplified maintenance therapy with ATV and RTV alone after virologic suppression does not markedly increase the risk of virologic failure.

DETAILED DESCRIPTION:
The expense, difficulty, and long-term adverse events associated with sustained adherence to combination antiretroviral therapy emphasize the need for simpler, alternative treatment strategies for HIV infection. Studies have shown that single protease inhibitor (PI) maintenance therapy may provide sufficient virologic suppression while reducing the risk of nucleoside reverse transcriptase inhibitor (NRTI)-associated metabolic complications. However, it is not known whether ritonavir-boosted atazanavir (ATV/RTV) maintenance therapy would be effective in controlling HIV replication in the genital compartments and whether viral load testing by blood collection would be effective in detecting elevated levels of HIV in the genital compartments. This study will determine whether simplified maintenance therapy with ATV/RTV after 48-week virologic suppression will increase the likelihood of virologic failure.

This study will last 54 weeks. Participants will undergo an electrocardiogram (EKG) at screening. At study start, participants will switch from their current PIs to ATV/RTV and stay on their current NRTIs until Week 6, when they will discontinue their NRTIs and remain on a maintenance regimen of ATV/RTV alone for the duration of the study. Study visits will take place at Weeks 3 and 6, then every 4 weeks until Week 30, then every 8 weeks until the end of the study at Week 54. Medication assessment, physical exam, and blood work will occur at each study visit. At Week 30, viral load will be measured in the genital secretions of both male and female study participants.

ELIGIBILITY:
Inclusion Criteria:

* HIV infected
* On first antiretroviral regimen, including at least 2 NRTIs and 1 PI, for at least 48 weeks immediately prior to study entry
* CD4 count of 250 cells/mm3 or greater
* Viral load less than 50 copies/ml within 30 days prior to entry
* Willing to use acceptable methods of contraception

Exclusion Criteria:

* Current or prior use of an NNRTI
* Certain PI mutations
* Hepatitis B infection within 90 days prior to study entry
* Certain therapies or medications within 30 days prior to study entry
* Heartbeat abnormalities or symptoms potentially related to heart block, such as unexplained fainting, dizziness, or palpitations, occurring within 180 days prior to study entry
* Drug or alcohol use or dependence that would interfere with adherence to the study requirements
* Serious illness requiring systemic treatment or hospitalization until the participant either completes therapy or has been clinically stable on therapy for at least 14 days prior to study entry
* Allergy or sensitivity to study medications or their formulations
* Current involuntarily incarceration for treatment of either a mental or physical illness
* Treatment for an active AIDS-defining opportunistic infection within 30 days prior to screening
* Pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2004-07; Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
Virologic failure, defined as 2 consecutive viral load measurements of 200 copies/ml or greater, at or before Week 30 (24 weeks on ATV/RTV alone)

SECONDARY OUTCOMES:
Grade 3 and 4 laboratory abnormalities and signs and symptoms
time to treatment discontinuation because of toxicity or intolerance
virologic failure at or before Week 54
viral load determined by modified ultrasensitive RT-PCR assay
minor PI variants at virologic failure
total cholesterol, high-density lipoprotein (HDL) cholesterol, calculated low-density lipoprotein (LDL) cholesterol, and triglycerides
CD4 cell count and percentages at Weeks 30 and 54
self-reported adherence scores
plasma drug levels characterized by Cmin and AUC
detectable viral load in the genital compartment at Week 30

CONTACTS AND LOCATIONS:
Overall Officials: Susan Swindells, MD, Study Chair — University of Nebraska
Locations (12):
- United States (11):
  - Stanford AIDS Clinical Trials Unit CRS, Palo Alto, California
  - University of Colorado Hospital CRS, Aurora, Colorado
  - Univ. of Hawaii at Manoa, Leahi Hosp., Honolulu, Hawaii
  - Univ. of Iowa Healthcare, Div. of Infectious Diseases, Iowa City, Iowa
  - Univ. of Nebraska Med. Ctr., Durham Outpatient Ctr., Omaha, Nebraska
  - Weill Cornell Chelsea CRS, New York, New York
  - Chapel Hill CRS, Chapel Hill, North Carolina
  - Duke Univ. Med. Ctr. Adult CRS, Durham, North Carolina
  - Cincinnati CRS, Cincinnati, Ohio
  - University of Pittsburgh CRS, Pittsburgh, Pennsylvania
  - Dallas VAMC, Dallas, Texas
- Puerto Rico AIDS Clinical Trials Unit CRS, San Juan, Puerto Rico

REFERENCES:
- [Background] Havlir DV, Marschner IC, Hirsch MS, Collier AC, Tebas P, Bassett RL, Ioannidis JP, Holohan MK, Leavitt R, Boone G, Richman DD. Maintenance antiretroviral therapies in HIV-infected subjects with undetectable plasma HIV RNA after triple-drug therapy. AIDS Clinical Trials Group Study 343 Team. N Engl J Med. 1998 Oct 29;339(18):1261-8. doi: 10.1056/NEJM199810293391801. PMID 9791141
- [Background] Pialoux G, Raffi F, Brun-Vezinet F, Meiffredy V, Flandre P, Gastaut JA, Dellamonica P, Yeni P, Delfraissy JF, Aboulker JP. A randomized trial of three maintenance regimens given after three months of induction therapy with zidovudine, lamivudine, and indinavir in previously untreated HIV-1-infected patients. Trilege (Agence Nationale de Recherches sur le SIDA 072) Study Team. N Engl J Med. 1998 Oct 29;339(18):1269-76. doi: 10.1056/NEJM199810293391802. PMID 9791142
- [Background] Reijers MH, Weverling GJ, Jurriaans S, Wit FW, Weigel HM, Ten Kate RW, Mulder JW, Frissen PH, van Leeuwen R, Reiss P, Schuitemaker H, de Wolf F, Lange JM. Maintenance therapy after quadruple induction therapy in HIV-1 infected individuals: Amsterdam Duration of Antiretroviral Medication (ADAM) study. Lancet. 1998 Jul 18;352(9123):185-90. doi: 10.1016/s0140-6736(98)06193-5. PMID 9683207
- [Background] Kahlert C, Hupfer M, Wagels T, Bueche D, Fierz W, Walker UA, Vernazza PL. Ritonavir boosted indinavir treatment as a simplified maintenance "mono"-therapy for HIV infection. AIDS. 2004 Apr 9;18(6):955-7. doi: 10.1097/00002030-200404090-00017. No abstract available. PMID 15060447
- [Background] Kelly M. Induction-maintenance antiretroviral strategies to reduce long-term toxicity. J HIV Ther. 2003 Feb;8(1):11-4. PMID 12840709
- [Result] Swindells S, DiRienzo AG, Wilkin T, Fletcher CV, Margolis DM, Thal GD, Godfrey C, Bastow B, Ray MG, Wang H, Coombs RW, McKinnon J, Mellors JW; AIDS Clinical Trials Group 5201 Study Team. Regimen simplification to atazanavir-ritonavir alone as maintenance antiretroviral therapy after sustained virologic suppression. JAMA. 2006 Aug 16;296(7):806-14. doi: 10.1001/jama.296.7.806. PMID 16905786
- [Derived] McKinnon JE, Mailliard RB, Swindells S, Wilkin TJ, Borowski L, Roper JM, Bastow B, Kearney M, Wiegand A, Mellors JW, Rinaldo CR; A5201 study team. Baseline natural killer and T cell populations correlation with virologic outcome after regimen simplification to atazanavir/ritonavir alone (ACTG 5201). PLoS One. 2014 May 6;9(5):e95524. doi: 10.1371/journal.pone.0095524. eCollection 2014. PMID 24802242
- [Derived] Wilkin TJ, McKinnon JE, DiRienzo AG, Mollan K, Fletcher CV, Margolis DM, Bastow B, Thal G, Woodward W, Godfrey C, Wiegand A, Maldarelli F, Palmer S, Coffin JM, Mellors JW, Swindells S. Regimen simplification to atazanavir-ritonavir alone as maintenance antiretroviral therapy: final 48-week clinical and virologic outcomes. J Infect Dis. 2009 Mar 15;199(6):866-71. doi: 10.1086/597119. PMID 19191590